CLINICAL TRIAL: NCT03131739
Title: Alaska Native Resilience Research Study
Brief Title: Alaska Native Collaborative Hub for Resilience Research
Acronym: ANCHRR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Alaska Fairbanks (Other)
Collaborators: University of Massachusetts, Amherst (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Stacy Rasmus, Research Associate Professor, University of Alaska Fairbanks
Other Study IDs: U19MH113138-01 (NIH)
Record Dates: First submitted 2017-04-18; First posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Suicide
Keywords: Resilience; Alaska Native; Community Based Participatory Research; Culture and Community Factors; Protective Factors; Risk Factors
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Community Level Assessment: 65 communities will undergo assessment of community / structural variables through review of public records and 3-5 key community interviewees per community.
- Individual Level Assessment: A subset of 6 communities will be elected through a stratification process. Youth will complete a set of protective factors measures and outcomes. Adults will complete a section of the Neighborhood Matters survey.

SUMMARY:
The goal of the Alaska Native Resilience Research Study (ANRRS) is to identify community-level protective factors that can most effectively reduce co-occurring youth suicide and alcohol risk. The following specific aims will help us achieve this overarching goal. The research team will: (1): Assess the association of a set of modifiable cultural, community and institutional factors (protective community factors) with suicide, suicidal behaviors (ideation, attempt), and associated adverse outcomes (accidental death, alcohol-misuse requiring healthcare) in 64 rural and remote Alaska Native villages to identify community-level factors that are most predictive of youth health outcomes; (2): In a stratified random sample of six communities, use quantitative methods to test a multi-level model of individual-level youth protective factors as predictors of individual-level youth resilience from suicide risk outcomes; and (3): Develop and disseminate a method-Alaska Community Resilience Mapping (AK-CRM)-for communities to measure and strategically strengthen their protective capabilities to increase youth health and reduce the risk for suicide.

Methodology:

DETAILED DESCRIPTION:
The ANCHRR builds on our established tribal partnerships in the three regions of Alaska with the highest need for effective, culturally congruent and community-based suicide prevention. Drs. Rasmus and Allen have been working collaboratively with Yup'ik communities in the Yukon Kuskokwim region and Dr. Wexler has been doing community-based participatory research in Northwest Alaska (NWA) for 20 years. Both research teams have spent this time partnering with tribal communities and developing evidence-based and self-determined suicide prevention initiatives that reflect local, AN understandings and values, strengthen community systems of support, and build local capacity for strategic prevention practice. The collaborative hub will extend this successful partnership model to include all of the tribal health regions across the state. With relevance for all of rural Alaska, the Alaska Native Resilience Study will provide important insights into the community level factors-institutions, traditions, resources and leaders-and mechanisms-the community perceptions, practices and norms-that increase resilience from suicide and reduce risk. The resulting Alaska Community Resilience Mapping (AK-CRM) Tool will provide a user-friendly, visual representation of the community-level protective factors and processes, and will engage Alaska community members in identifying the community-level protective factors in their community and will offer scientifically-based recommendations for action. In this way, ANCHRR's proposed activities translate results from the research study into practical suggestions for tribal leaders, local practitioners and policy makers, to maximize its public health impact.

ELIGIBILITY:
Inclusion Criteria:

* To identify persons able to assess diverse community protective factors, we will identify at least 5 village members from each community who are: (a) local school board members or school workers, (b) community health aids, (c) village-based counselors, (d) tribal council members or tribal administrators, (e) city managers, (f) village public safety officers or village public officers, (g) postmasters, (h) Elder council members, and/or (i) religious leaders. This initial village list will also include other people who are informal leaders in the village.

Exclusion: From this list, participants will be screened to ensure: (1) village residence or service provision in the community for at least 5 years cumulatively and (2) endorsements from members of the Research Steering Committee, who are knowledgeable about specific community dynamics.

* The sample of 64 communities will be stratified into higher, medium and lower protection community groups using their protective community factor score from Aim 1, then 6 communities will be randomly selected, 2 from each stratification group.
* Children in each of 6 selected communities
* All adults 18-29 in 6 selected communities.
* Approximately 15 individual adults will be recruited in each of the six villages (n=60) through sampling the following sectors of community: government, church, social service, store/business, school, health care, parent, elder. We will contact individuals nominated in each sector by the local tribal council or their designate.

Exclusion Criteria:

* Communities with fewer than 150 people will be excluded since the protective community dynamics and adverse outcomes are more stable in larger villages. This reduces the number of participating communities from 71 total number of villages to 65.
* We will exclude children under the age of 15, because we seek information regarding late adolescence and beginning adulthood. We will exclude children who do not have the capacity to assent or to participate in the computerized survey.
* We will exclude adults who do not have the capacity to consent or to participate in the computerized survey.
* We will exclude adults who have lived in their respective village for less than 5 years, because we will be asking for information about community factors that require perspectives over time. We will exclude adults who do not have the capacity to consent or to participate in the computerized survey.

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Sixty-five Alaska Native communities (villages) will be drawn from a regional sample and individual study participants will be drawn from a community sample consisting of six Alaska Native villages across three regions.
Sampling Method: Non-Probability Sample
Enrollment: 585 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Community Level Assessment: suicide and accidental deaths | Year 2
  The Trauma Registry and the Alaska Violent Death Reporting System (AKVDRS) will be used to document suicide and accidental deaths

SECONDARY OUTCOMES:
Individual Level Assessment: Youth: Individual: Communal Mastery Scale | Year 4
  Collective efficacy: solving life challenges through joining with others
Individual Level Assessment: Youth: Family: Family Relationship Scale | Year 4
  Quality of family relationships
Individual Level Assessment: Suicide Risk Resilience: Reasons for Life | Year 4
  Alaska Native cultural beliefs and experiences that make life enjoyable, worthwhile, and provide meaning
Community Level Assessment: Community Protective Factors | Year 2
  A structured interview guide will ask community experts in each village about the extent to which protective factors related to effective services, community development, self-determination/local control, cultural continuity are present
Individual Level Assessment: Alcohol Risk: Reflective Processes Resilience: Reflective Processes | Year 4
  9-item measure of awareness of the reciprocal consequences of one's behavior across people and time, and focuses on reasons for sobriety through a culturally patterned type of awareness used in thinking over potential negative consequences of alcohol
Individual Level Assessment: Youth: Community: Community Protective Factors | Year 4
  Perceived support and opportunities in community
Individual Level Assessment: Youth: Social Connection: Awareness of Connectedness | Year 4
  Awareness of the interrelated welfare of the individual with family, community, and the natural environment
Individual Level Assessment: Adult: Protective Community Factors: Protective Community Factors | Year 4
  Community level organizational features of local control and cultural continuity
Individual Level Assessment: Adult: Community Social Processes: Informal Social Control | Year 4
  Question stem for generally held beliefs was, "People in this village believe that…" 6-items related to child welfare ("adults should know where their children are.", 10 items for child management ("adults should do something if a child is doing something dangerous"), 4-items related to adolescent behavior ("It is wrong for teenagers to fist fight."), 6-items related to crime ("People should do something if a neighbor's house is being vandalized.") and 5 items related to community member responsibility ("People should take action to make the village better.")

IPD SHARING:
Plan to Share IPD: Yes
The Tribal Health Organizations and the research team jointly own all data, consistent with the principles of community-based participatory research (CBPR). De-identified data and results will be shared at every meeting of the AN External Advisory Council, Collaborative Hub and Research Steering Committee. Datasets are shared by request and approval by the Tribal Health Organizations and Project PIs as they become available. The research team propose to development Tribal Data Sharing and Ownership Agreements (DSOA) with the three participating Tribal Health Organizations in Year 1 of the ANCHRR project.